CLINICAL TRIAL: NCT05517694
Title: Effect of Respiratory Exercises Applied In Addition to Pelvic Floor Exercises and Behavioral Therapy Methods on the Intravaginal Ejaculation Latency Time In Individuals With Premature Ejaculation Patients
Brief Title: Effect of Respiratory Exercises On The Intravaginal Ejaculation Latency Time
Acronym: premature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Dilber Karagozoglu Coskunsu, principal investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BahcesehirUn.
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Premature Ejaculation
Keywords: premature ejaculation; respiratory exercises; pelvic floor muscles endurance; pelvic floor muscles strength; parasympathetic activity; behavioral therapy
MeSH Terms: conditions — Premature Ejaculation | interventions — Behavior Therapy; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: 62 participants will randomly divided into two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be double blind (both participants and assessor blinded)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic floor exercises, behavioral therapy and respiratory exercises group (Experimental): Interventions of this group include pelvic floor exercises and behavioral therapy plus respiratory exercises for 8 weeks.
  Interventions: Other: Pelvic floor exercises and behavioral therapy; Other: Respiratory exercises
- pelvic floor exercises and behavioral therapy group (Active Comparator): Interventions of this group include pelvic floor exercises and behavioral therapy for 8 weeks.
  Interventions: Other: Pelvic floor exercises and behavioral therapy

INTERVENTIONS:
Other: Pelvic floor exercises and behavioral therapy — Pelvic floor exercises and behavioral therapy interventions include a 4-step treatment protocol: 1) awareness of the pelvic floor muscles, 2) teaching the specific contraction of the pelvic floor muscles, 3) teaching the timing of the contraction and maintenance of the pelvic floor muscles during the intercourse pre-orgasmic sensation with start-stop behavioral therapy, 4) the strengthening exercises of the pelvic floor muscles. For slow twitch fibers, 15 repetitive exercises including 10 seconds of submaximal contraction followed by 10 seconds of relaxation, and 10 repetitive exercises including 1 second submaximal contraction followed by 1 second relaxation for fast-twitch fibers will be given 2 times a day, 3 days a week, 8 weeks.
Other: Respiratory exercises — Pelvic floor exercises and behavioral therapy interventions include a 4-step treatment protocol: 1) awareness of the pelvic floor muscles, 2) teaching the specific contraction of the pelvic floor muscles, 3) teaching the timing of the contraction and maintenance of the pelvic floor muscles during the intercourse pre-orgasmic sensation with start-stop behavioral therapy, 4) the strengthening exercises of the pelvic floor muscles. For slow twitch fibers, 15 repetitive exercises including 10 seconds of submaximal contraction followed by 10 seconds of relaxation, and 10 repetitive exercises including 1 second submaximal contraction followed by 1 second relaxation for fast-twitch fibers will be given 2 times a day, 3 days a week, 8 weeks.
  Respiratory exercises will be given 6 breaths/minute with expiration and inspiration times of 7 seconds and 3 seconds, respectively. At least 10 diaphragmatic breaths will be given in each session, 2 times a day, 7 days a week, 8 weeks.
  Arms: pelvic floor exercises, behavioral therapy and respiratory exercises group

SUMMARY:
According to recent epidemiological studies, premature ejaculation (PE) is accepted as the most common sexual dysfunction in men, with a frequency of up to 20%.According to the definition made by the International Society for Sexual Medicine (ISSM) in 2014, PE: 'Ejaculation (lifelong PE) that is always or almost always around 1 minute after the first sexual experience, or, ejaculation time can be reduced to 3 minutes.

Male pelvic floor muscle function also plays a role in coordinating ejaculation. Pelvic floor therapy has been found to improve control over ejaculation and increase intravaginal ejaculatory delay times (IELT) in men with premature ejaculation and pelvic floor muscle dysfunction.

Behavioral treatments consist of physical techniques that will help men's sexual development, delaying ejaculation and increasing sexual self-confidence. Specific physical techniques include: The "stop-start" technique developed by Semans involves the person or their partner, the penis is stimulated until you feel the urge to ejaculate, then it stops until the feeling goes away and the feeling goes away; this is repeated several times before allowing ejaculation to occur.

The pelvic floor muscles have respiratory functions, and most of them have been investigated in studies on urological diseases. Focusing on lower abdominal respiration, it was observed that it was associated with a significant increase in whole blood serotonin 5-hydroxytryptamine (5-HT) levels . One hypothesis proposed for the pathophysiology of premature ejaculation is that high 5-HT is associated with ejaculatory control.

Our purpose is to investigate the effect of adding breathing exercises in addition to pelvic floor rehabilitation and behavioral treatment methods on ejaculation time in individuals with premature ejaculation.

DETAILED DESCRIPTION:
INTRODUCTION According to recent epidemiological studies, premature ejaculation (PE) is accepted as the most common sexual dysfunction in men, with a frequency of up to 20%. According to the definition made by the International Society for Sexual Medicine (ISSM) in 2014, PE: 'Ejaculation (lifelong PE) that is always or almost always around 1 minute after the first sexual experience, or, ejaculation time can be reduced to 3 minutes. A male sexual dysfunction characterized by clinically significant and bothersome shortening (acquired PE) up to and including an inability to always or almost always delay ejaculation at vaginal penetrations, and negative personal problems such as stress, distress, frustration, and/or sexual avoidance.

Ejaculation is a highly complex process that requires the coordination and efferent nerve interaction of the motor and sensory areas of the brain and spinal motor areas, as well as sensory receptors and afferent nerve pathways. Ejaculation is controlled by various neurotransmitters distributed throughout the supraspinal and spinal nuclei. In animal studies, serotonin [5-hydroxytryptophan (5-HT)], dopamine (DA) and oxytocin (OT), opioids, gamma aminobutyric acid (GABA), nitric oxide (NO) and norepinephrine (NE); GABA, OT, 5-HT and Substance P at the spinal cord level; Peripheral NE, acetylcholine (Ach), NO, OT, purines (P2), 5-HT and sensory receptors have been shown to be involved in ejaculation.

Despite pelvic floor physiotherapy, which represents a conservative, modifiable, non-invasive, non-pharmacological and non-surgical intervention in the treatment of male sexual dysfunction, the biological relationship between pelvic floor function and male sexual function is rarely emphasized.

Male pelvic floor dysfunction has been associated with ejaculation and orgasm dysfunction as well as erectile dysfunction. Male pelvic floor muscle function also plays a role in coordinating ejaculation. Pelvic floor therapy has been found to improve control over ejaculation and increase intravaginal ejaculatory delay times (IELT) in men with premature ejaculation and pelvic floor muscle dysfunction.

Behavioral treatments consist of physical techniques that will help men's sexual development, delaying ejaculation and increasing sexual self-confidence. Specific physical techniques include: The "stop-start" technique developed by Semans involves the person or their partner, the penis is stimulated until you feel the urge to ejaculate, then it stops until the feeling goes away and the feeling goes away; this is repeated several times before allowing ejaculation to occur. The goal is to learn and recognize feelings of arousal and to improve control over ejaculation. The "squeeze" technique proposed by Masters and Johnson, stimulates the penis until you feel the urge to ejaculate, then tightens the glans penis until the urge to ejaculate passes; this is repeated without allowing ejaculation to occur.

The pelvic floor muscles have respiratory functions, and most of them have been investigated in studies on urological diseases. Focusing on lower abdominal respiration, it was observed that it was associated with a significant increase in whole blood serotonin 5-hydroxytryptamine (5-HT) levels. One hypothesis proposed for the pathophysiology of premature ejaculation is that high 5-HT is associated with ejaculatory control. Psychological comorbidities such as depression, anxiety, and extreme stress are associated with premature ejaculation. It has been observed that pelvic and perineal muscles that have not been fully relaxed may cause premature ejaculation.

PURPOSE To investigate the effect of adding breathing exercises in addition to pelvic floor rehabilitation and behavioral treatment methods on ejaculation time in individuals with premature ejaculation.

METHOD 62 individuals between the ages of 18-45 with premature ejaculation problems will be included in the study. Participating in the study will be randomly divided into two groups. To the 1st group (n=32), 1) awareness of the pelvic floor muscles, 2) teaching the specific contraction of the pelvic floor muscles, 3) teaching the timing of the contraction and maintenance of the pelvic floor muscles during the intercourse pre-orgasmic sensation with start stop technique, 4) the strengthening exercises of the pelvic floor muscles. A 4-step treatment protocol will be applied. Pelvic floor muscle strengthening exercises will be given for both slow-twitch and fast-twitch fibers. For slow twitch fibers, 15 repetitive exercises including 10 seconds of submaximal contraction followed by 10 seconds of relaxation, and 10 repetitive exercises including 1 second submaximal contraction followed by 1 second relaxation for fast-twitch fibers will be given 2 times a day, 3 days a week. Slow and fast twitch fiber contraction exercises will require maximum contraction of the specific pelvic floor muscles without contraction of the gluteal and abdominal and adductor muscles. In the second group (n=32), breathing exercises will be given in addition to this treatment protocol. Diaphragmatic breathing exercises will be given 6 breaths/minute, expiration and inspiration times of 7 seconds and 3 seconds, respectively, and at least 10 diaphragmatic breaths will be given in each session, 3 times a day, 8 weeks. All individuals to be included in the study will be selected, according to The International Society for Sexual Medicine (ISSM), who always or almost always ejaculate 1 minute or more before vaginal penetration. Intravaginal ejaculation time (IELT) will be evaluated for both groups before and after the application. Before the application, pelvic floor muscle strength and endurance of both groups will be evaluated by ultrasound.

Inclusion criteria for the study:

* IELT < 60 seconds
* PEDT > 11
* Persons included in the study have been in a stable relationship with a partner for at least 6 months and have sexual intercourse once a week or more

Exclusion criteria from the study:

* Individuals with erectile dysfunction
* Individuals with prostatitis
* Those who have a psychiatric disorder and take medication for this reason

ELIGIBILITY:
Inclusion Criteria:

* IELT < 60 seconds
* PEDT > 11
* Persons included in the study have been in a stable relationship with a partner for at least 6 months and have sexual intercourse once a week or more

Exclusion Criteria:

* Individuals with erectile dysfunction
* Individuals with prostatitis
* Those who have a psychiatric disorder and take medication for this reason

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Intravaginal Ejaculatation Latency Time(IELT) | Change from pre-treatment of Intravaginal Ejaculatory Latency Time and at the end of the 8 weeks after treatment.
  Intravaginal ejaculation latency time (IELT) is the time it takes to ejaculate during vaginal penetration. An intravaginal ejaculation time if less than 1 minute is defined as premature ejaculation.

SECONDARY OUTCOMES:
Pelvic Floor Muscles Contraction and Endurance Assesment | Change from pre-treatment of pelvic floor contraction and endurance with ultrasound and at the end of the 8 weeks after treatment.
  Pelvic floor muscle contraction will be done by measuring with ultrasound the amount of bladder floor movement. 1 hour before the test, all participants will be asked to fill their bladders by consuming 600-750 ml of water within half an hour without urinating.
Assessment of the Autonomic Nervous System | Change from pre-treatment of autonomic nervous system data from elite hrv device and at the end of the 8 weeks after treatment.
  Elite HRV device will attached to the index fingers of the patients in the sitting position, and data is collected and recorded for 1 minute. The expression RMSSD is used for a snapshot of the Parasympathetic branch of the Autonomic Nervous System and is the basis for your HRV score. PNN50 refers to NN50 divided by the total number of NN (R-R) intervals. NN50 is the number of consecutive pairs of NN (R-R) intervals that differ by more than 50 ms (Heathers, 2014). LF power is the efficiency of the frequency in the range of 0.04 - 0.15 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Ümit Erkut, PhD(c),PT, Principal Investigator — Bahçeşehir University; Dilber Karagozoglu Coskunsu, PhD,PT, Study Chair — Fernerbahce University; Ali Veysel Ozden, PhD,MD, Study Chair — Bahçeşehir University; Kubra Erkut, PT, Study Chair — Kurbaa Egitim Danısmanlık
Locations (1):
- Kurbaa Egitim Danısmanlık Merkezi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Porst H, Montorsi F, Rosen RC, Gaynor L, Grupe S, Alexander J. The Premature Ejaculation Prevalence and Attitudes (PEPA) survey: prevalence, comorbidities, and professional help-seeking. Eur Urol. 2007 Mar;51(3):816-23; discussion 824. doi: 10.1016/j.eururo.2006.07.004. Epub 2006 Jul 26. PMID 16934919
- [Result] Serefoglu EC, McMahon CG, Waldinger MD, Althof SE, Shindel A, Adaikan G, Becher EF, Dean J, Giuliano F, Hellstrom WJ, Giraldi A, Glina S, Incrocci L, Jannini E, McCabe M, Parish S, Rowland D, Segraves RT, Sharlip I, Torres LO. An evidence-based unified definition of lifelong and acquired premature ejaculation: report of the second International Society for Sexual Medicine Ad Hoc Committee for the Definition of Premature Ejaculation. J Sex Med. 2014 Jun;11(6):1423-41. doi: 10.1111/jsm.12524. Epub 2014 May 22. PMID 24848805
- [Result] Waldinger MD. Recent advances in the classification, neurobiology and treatment of premature ejaculation. Adv Psychosom Med. 2008;29:50-69. doi: 10.1159/000126624. PMID 18391557
- [Result] Gao J, Zhang X, Su P, Liu J, Xia L, Yang J, Shi K, Tang D, Hao Z, Zhou J, Liang C. Prevalence and factors associated with the complaint of premature ejaculation and the four premature ejaculation syndromes: a large observational study in China. J Sex Med. 2013 Jul;10(7):1874-81. doi: 10.1111/jsm.12180. Epub 2013 May 7. PMID 23651451
- [Result] McMahon CG, Jannini EA, Serefoglu EC, Hellstrom WJ. The pathophysiology of acquired premature ejaculation. Transl Androl Urol. 2016 Aug;5(4):434-49. doi: 10.21037/tau.2016.07.06. PMID 27652216
- [Result] Corona G, Rastrelli G, Limoncin E, Sforza A, Jannini EA, Maggi M. Interplay Between Premature Ejaculation and Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2015 Dec;12(12):2291-300. doi: 10.1111/jsm.13041. Epub 2015 Nov 9. PMID 26552599